CLINICAL TRIAL: NCT06329908
Title: Single-arm, Open, Prospective Clinical Study of Neoantigen-loaded Dendritic Cell Vaccine (Neo-DCVac) Combined With Immune Checkpoint Inhibitors (ICIs) in the Treatment of Advanced Lung Cancer Resistant to ICIs
Brief Title: DC Combined With ICIs in the Treatment of Advanced Lung Cancer Resistant to ICIs
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhen-Yu Ding (Other)
Responsible Party: Sponsor-Investigator, Zhen-Yu Ding, Clinical Professor, Sichuan University
Organization: Sichuan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSLG-001
Record Dates: First submitted 2023-12-28; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer
Keywords: Criteria for inclusion
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- (Neo-DCVac) combined with immune checkpoint inhibitors (ICIs) (Experimental): DC cell injection ,1.5 × 10 7/time, subcutaneous multi-point injection in axilla and groin or lymph node injection guided by color Doppler ultrasound in axilla and groin, continuous injection at 0W, 1W, 3W, 5W and 7W for five times as the first immunization cycle. Tumor response was evaluated 2 weeks after the completion of the first immunotherapy cycle, and treatment was continued if the response was evaluated as effective (SD/PR/CR), and every 3 weeks until disease progression or intolerable toxicity or active withdrawal of the patient, whichever came first.ICIs are PD1/PD-L1 inhibitors and continue to be pre-enrollment ICIs of any brand
  Interventions: Drug: LG002

INTERVENTIONS:
Drug: LG002 — Neo-DCVac combined with ICIs in the treatment of advanced lung cancer resistant to ICIs.
  Other Names: ICIs

SUMMARY:
This is a single-center, single-arm, prospective clinical trial to investigate the safety and efficacy of Neo-DCVac combined with ICIs in the treatment of advanced lung cancer resistant to ICIs.

DETAILED DESCRIPTION:
The study screened patients with PD-1 immunochemotherapy in the first-line treatment regimen, and extracted tumor tissues from patients after PD-1 resistance for neoantigen prediction. During neoantigen screening and vaccine preparation, patients received a second-line regimen (docetaxel) as bridging therapy. After completion of bridging therapy and the patient 's vaccine preparation was successful, the patient started receiving the vaccine combined with ICIs. The completion of 5 vaccine injections was followed by an immunization course. Efficacy was assessed 2 weeks after the end of an immunization course, and if effective (tumor response evaluated as SD/PR/CR), the next cycle of immunotherapy was continued, with subsequent treatments administered every 3 weeks until disease progression or severe intolerance occurred or the patient requested withdrawal, whichever came first.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-85 years.
* ECOG score was 0-2.
* Histological or cytological diagnosis confirmed non-small cell lung cancer, which was staged IIIB-IV according to AJCC version 8.
* Patients have received first-line chemotherapy combined with ICIs (PD1/PD-L1, ICIs type is not limited) and developed drug resistance.
* Normal function of major organs, that is, meeting the following criteria: a) blood routine examination (hematopoietic growth factors and blood transfusion were not used within 7 days): granulocyte count ≥ 1.5 × 109/L, platelet count ≥ 80 × 109/L, hemoglobin ≥ 80 g/L; b) biochemical examination: total bilirubin ≤ 1.5 × ULN (upper limit of normal); serum alanine aminotransferase (ALT) or serum aspartate aminotransferase (AST) ≤ 2.5 × ULN; creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula); c) coagulation function: INR or PT ≤ 1.5 × ULN (upper limit of normal), if the subject is receiving anticoagulant therapy, as long as PT is in the range proposed by anticoagulant drugs; d) urine routine examination: urine routine examination urine protein ≥ 2 +, 24-hour urine protein quantitative examination should be performed, such as quantitative urine protein ≤ 1 g/24 h.
* Female subjects of childbearing age or male subjects with sexual partners of childbearing age should take effective contraceptive measures throughout the treatment period and 6 months before and after the treatment period.
* Subjects voluntarily participate in the study and sign the informed consent form

Exclusion Criteria:

* The pathological type is mixed type, containing small cell carcinoma or other types of components.
* with the blood-borne infectious disease HIV.
* History of mental disorder, drug abuse and drug abuse.
* Any other malignancy (except completely cured cervical carcinoma in situ or basal cell or squamous cell skin cancer) within 3 years.
* Accompanied by other immune diseases, or long-term use of immunosuppressive agents or hormones.
* Any unstable systemic disease (including active uncontrolled gastrointestinal ulcers, gastric obstruction, bleeding risk or coagulopathy, active infection, for subjects with hepatitis B, anti-hepatitis B 11 virus treatment is required during study treatment, active hepatitis C subjects (HCV antibody positive and HCV- RNA levels above the lower limit of detection, grade IV hypertension, unstable angina pectoris, congestive heart failure, myocarditis, unstable cerebrovascular disease, thrombotic disease, liver, kidney, uncontrolled metabolic disease or unhealed fractures, wounds as judged by the surgeon).
* Presence of active central nervous system (CNS) metastases; subjects with previously treated brain metastases (e.g., surgery, radiotherapy, hormone therapy) are allowed if clinically stable for at least two weeks after treatment from the first dose of study drug and corticosteroids are discontinued 7 days before study drug administration; untreated, asymptomatic subjects with brain metastases (i.e., no neurological symptoms, no need for corticosteroids, no significant edema around the brain metastases) can be enrolled.
* Any anti-tumor therapy including chemotherapy, radiotherapy, and targeted therapy within 3 weeks prior to the first dose of study drug.
* Presence of pleural effusion, pericardial effusion, or ascites with clinical symptoms or requiring drainage.
* Previous use of anti-tumor vaccines, live vaccines within 30 days.
* Patients are difficult to communicate or to follow up for a long time. Pregnant or lactating women.
* Current or planned participation in other clinical trials.
* Dr. finds other unsuitable situations

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
The safety of Neo-DCVac combined with ICIs. | 2 years
  This study will collected any adverse medical events that occurred during the study drug treatment, and the treatment-related adverse events as assessed by" CTCAE v5.0".

SECONDARY OUTCOMES:
The efficacy of Neo-DCVac combined with ICIs. | 2 years
  Using the revisit1.1 tumor evaluation criteria for efficacy evaluation, evaluate disease progression free survival (PFS) .
The efficacy of Neo-DCVac combined with ICIs. | 2 years
  Using the revisit1.1 tumor evaluation criteria for efficacy evaluation, evaluate disease objective response rate (ORR).

OTHER OUTCOMES:
Synergistic anti-tumor mechanism. | 2 years
  The immune response of subjects was assessed by peripheral blood cell flow cytometry within 2 weeks after the initial immunotherapy and every 3 months during the immunomaintenance treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Li, MD, Study Chair — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No